CLINICAL TRIAL: NCT07099677
Title: The Effect of Antihypertensive Medication Use on Fall Risk: A Randomized Controlled Trial
Brief Title: Short-Term Effects of Antihypertensive Drugs on Postural Balance and Fall Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Alp Ozel, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-AO-05
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypertension; Fall Risk; Postural Balance; Fear of Falling
Keywords: Antihypertensive drugs; Fall risk; Hypertension; Medication-related falls; Postural balance; Randomized controlled trial
MeSH Terms: conditions — Hypertension | interventions — Adrenergic beta-Antagonists; Angiotensin-Converting Enzyme Inhibitors; Calcium Channel Blockers

STUDY DESIGN:
Intervention Model Description: Participants diagnosed with primary hypertension will be randomly assigned to one of three parallel treatment groups using block randomization: beta-blocker (e.g., Metoprolol), ACE inhibitor (e.g., Ramipril), or calcium channel blocker (e.g., Amlodipine). Each group will receive its assigned intervention independently and concurrently, and outcome measures will be assessed at baseline, week 2, and week 4.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participants and the outcomes assessors will be masked to group allocation. Participants will not be informed about the specific antihypertensive drug they receive, and the individuals conducting the balance and symptom assessments will remain blinded to the treatment groups to reduce assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beta Blocker Group (Experimental): Participants will receive a beta blocker (e.g., Metoprolol) for antihypertensive treatment.
  Interventions: Drug: Beta Blocker
- ACE Inhibitor Group (Experimental): Participants will receive an ACE inhibitor (e.g., Ramipril) for antihypertensive treatment.
  Interventions: Drug: ACE inhibitor
- Calcium Channel Blocker Group (Experimental): Participants will receive a calcium channel blocker (e.g., Amlodipine) for antihypertensive treatment.
  Interventions: Drug: Calcium channel blocker

INTERVENTIONS:
Drug: Beta Blocker — Participants in this group will receive standard antihypertensive treatment with a beta-adrenergic receptor blocker. The exact agent and dosage will be determined by the cardiology clinic according to clinical guidelines. Balance and fall risk assessments will be conducted at baseline (T0), week 2 (T1), and week 4 (T2).
  Other Names: Beta-Adrenergic Receptor Blocker; β-blocker; Beta-adrenergic antagonist
  Arms: Beta Blocker Group
Drug: ACE inhibitor — Participants in this group will receive standard antihypertensive treatment with an angiotensin-converting enzyme inhibitor. The dose and specific agent will be prescribed based on routine clinical criteria. Assessments will take place at T0, T1, and T2.
  Other Names: Angiotensin-converting enzyme blocker; ACEI; Standard ACE inhibitor therapy
  Arms: ACE Inhibitor Group
Drug: Calcium channel blocker — This group will receive a calcium channel blocker as part of their standard hypertension management. Dosage and agent will follow standard cardiology practice. Postural balance and fall risk will be measured at all study time points.
  Other Names: Calcium Antagonist; CCB; Standard CCB therapy
  Arms: Calcium Channel Blocker Group

SUMMARY:
The goal of this clinical trial is to compare the short-term effects of three commonly prescribed antihypertensive drug classes (beta-blockers, ACE inhibitors, and calcium channel blockers) on postural balance and fall risk in adults with newly diagnosed primary hypertension. The main questions it aims to answer are:

* Do different antihypertensive drugs affect objective balance performance and fall risk?
* What are the effects of these medications on dizziness and fear of falling?

Researchers will use a balance analysis system (Biodex Balance System) and self-reported scales (Dizziness Handicap Inventory and Falls Efficacy Scale) to assess outcomes. Participants will:

* Be randomly assigned to one of three drug groups (metoprolol, ramipril, or amlodipine)
* Be evaluated at baseline (prior to treatment), at 2 weeks, and at 4 weeks after starting treatment
* Complete balance tests and questionnaires at each time point

This study aims to provide clinical insight into how commonly used blood pressure medications may impact balance and fall risk in real-world settings.

DETAILED DESCRIPTION:
Falls and balance impairments are significant health concerns, particularly in individuals with hypertension who may be starting pharmacological treatment. Some antihypertensive drugs are known to cause side effects such as dizziness, postural hypotension, and impaired balance, all of which can increase fall risk. Despite this, comparative evidence on the short-term impact of different antihypertensive drug classes on postural balance remains limited.

This randomized controlled trial aims to compare the effects of three first-line antihypertensive drug classes-beta-blockers (e.g., metoprolol), ACE inhibitors (e.g., ramipril), and calcium channel blockers (e.g., amlodipine)-on postural stability and fall risk during the initial four weeks of treatment. Participants will be individuals aged 18-75 years who have been newly diagnosed with primary hypertension and have not previously used antihypertensive medications.

Assessments will be conducted using both objective and subjective measures. Objective balance evaluations will be performed using the Biodex Balance System, including the Fall Risk Test, Postural Stability Test (overall, anterior-posterior, and medial-lateral stability indices), and the Clinical Test of Sensory Interaction on Balance (CTSIB). Subjective assessments will include the Falls Efficacy Scale (FES) to evaluate fear of falling and the Dizziness Handicap Inventory (DHI) to assess the impact of dizziness on daily life.

The trial will include three evaluation time points: baseline (before starting treatment), week 2, and week 4. By providing a multidimensional assessment of balance performance, the study seeks to identify potential safety concerns and guide clinicians in making informed treatment decisions based on both cardiovascular and postural health.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years
* Newly diagnosed with primary hypertension
* No prior use of antihypertensive medication
* No history of neurological, vestibular, orthopedic, or psychiatric conditions affecting balance
* Able to walk independently without assistive devices
* Provided written informed consent to participate in the study

Exclusion Criteria:

* Secondary hypertension
* Known diagnosis of vestibular disorders (e.g., BPPV, Ménière's disease)
* Use of medications that may affect balance (e.g., sedatives, psychotropic drugs)
* History of falls due to trauma unrelated to balance
* Cognitive impairment preventing proper test participation
* Inability to complete the assessments at follow-up timepoints (2nd and 4th week)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Fall Risk Score (Biodex Balance System) | Baseline (T0), Week 2 (T1), Week 4 (T2)
  Objective assessment of fall risk using the Fall Risk Test on the Biodex Balance System. Higher scores indicate greater fall risk.

SECONDARY OUTCOMES:
Postural Stability Indices (OSI, APSI, MLSI) | Baseline (T0), Week 2 (T1), Week 4 (T2)
  Stability scores reflecting anterior-posterior and medial-lateral sway during standing, measured by the Biodex Balance System.
Sensory Integration Scores (CTSIB) | Baseline (T0), Week 2 (T1), Week 4 (T2)
  Composite scores from the Clinical Test of Sensory Interaction on Balance, measuring sensory contributions to balance.
Falls Efficacy Scale (FES) Score | Baseline (T0), Week 2 (T1), Week 4 (T2)
  Self-reported fear of falling during daily activities, total score ranges from 10 to 40.
Dizziness Handicap Inventory (DHI) - Total and Subscale Scores | Baseline (T0), Week 2 (T1), Week 4 (T2)
  Measures physical, emotional, and functional impact of dizziness. Total score range: 0-100.

OTHER OUTCOMES:
Presence of Orthostatic Hypotension | Baseline (T0)
  Dichotomous variable assessed at baseline (T0). Binary (Yes/No)
Presence of Dizziness | Baseline (T0)
  Dichotomous variable assessed at baseline (T0). Binary (Yes/No).
Demographics (Age, BMI, Gender) | Baseline (T0)
  Baseline covariates used for subgroup and interaction analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ozel, PT, PhD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Izzet Baysal Training and Research Hospital, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the publication-including demographic variables, group allocation, balance test scores (Fall Risk Score, OSI, APSI, MLSI, CTSIB), Falls Efficacy Scale (FES), Dizziness Handicap Inventory (DHI) scores, and related clinical data (e.g., presence of orthostatic hypotension, reported dizziness)-will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting documents will be available starting after the main results are published in a peer-reviewed journal and will remain accessible indefinitely via the Zenodo repository (https://zenodo.org). A permanent DOI will be provided upon upload.
Access Criteria: Anyone may access the de-identified data without restriction via the digital object identifier (DOI) assigned at the time of publication.
URL: https://zenodo.org